CLINICAL TRIAL: NCT04965818
Title: A Phase 1b/2 Open-label, Nonrandomized Study of FGFR Inhibitor Futibatinib in Combination With MEK-inhibitor Binimetinib in Patients With Advanced KRAS Mutant Cancer
Brief Title: Phase 1b/2 Study of Futibatinib in Combination With Binimetinib in Patients With Advanced KRAS Mutant Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic decision by sponsor.
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAS-120-204
Record Dates: First submitted 2021-07-06; First posted 2021-07-16 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Advanced or Metastatic Solid Tumors Irrespective of Gene Alterations; Non-Small Cell Lung Cancer; KRAS Gene Mutation
Keywords: Futibatinib; Binimetinib; MEKi; FGFR; FGFRi; TAS-120; KRASmt; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — futibatinib; binimetinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Futibitanib in combination with binimetinib (Experimental): Dose escalation: Futibitanib in combination with binimetinib in patients with advanced cancer disease.
  Dose expansion: Futibatinib in combination with binimetinib at the RP2D in patients with advanced KRASmt NSCLC
  Interventions: Drug: Futibatinib and Binimetinib

INTERVENTIONS:
Drug: Futibatinib and Binimetinib — Patients will receive futibatinib once daily in combination with binimetinib twice daily by oral administration on a 21-day cycle

SUMMARY:
Phase 1b/2 study to evaluate the FGFRi futibatinib in combination with the MEKi binimetinib in patients with advanced KRASmt tumors.

DETAILED DESCRIPTION:
This is an open-label, nonrandomized, uncontrolled Phase 1b/2 study to determine the recommended phase 2 dose (RP2D) of futibatinib in combination with binimetinib and to explore the preliminary antitumor activity of futibatinib in combination with binimetinib in patients with advanced KRASmt tumors.

The study will consist of two parts:

* Part 1: Dose-Escalation part to determine the RP2D and dosing schedule of futibatinib in combination with binimetinib in patients with advanced cancer disease
* Part 2: Dose-Expansion part to evaluate the preliminary antitumor activity of futibatinib in combination with binimetinib at the RP2D in patients with advanced KRASmt NSCLC

Patients will receive study treatment until progressive disease or any other discontinuation or withdrawal criterion is met.

No patients were enrolled in Phase 2 as the Sponsor decided to not proceed with the dose expansion Phase 2 part of the TAS-120-204 study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced cancer of any tumor type (Part 1) or NSCLC with a confirmed KRAS mutation as determined by local results (Part 2)
* Appropriate candidate for experimental therapy
* For patients in Part 2 only: Patient has radiographically measurable disease per RECIST 1.1 criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Adequate cardiac function (Left ventricular ejection fraction (LVEF) ≥50% )
* Adequate organ function
* Must have tumor tissue specimen available (optional for patients in Part 1)

Exclusion Criteria:

* History or current evidence of calcium and phosphate hemostasis disorder or systemic mineral imbalance with ectopic calcification of soft tissues
* Current evidence or history of clinically significant corneal or retinal disorder as confirmed by ophthalmologic examination.
* Known untreated central nervous system (CNS) metastases or history of uncontrolled seizures.
* Significant gastrointestinal disorder(s) that could interfere with absorption of futibatinib/binimetinib
* Patients who have neuromuscular disorders that are associated with elevated creatinine kinase (CK)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2023-06-11 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) in Part 1 | 12 months
  Determine RP2D of futibatinib in combination with binimetinib based on Dose Limiting Toxicities
Objective Response Rate (ORR) in Part 2 | approximately 24 months
  proportion of patients who have achieved a PR or complete response (CR) according to RECIST 1.1.

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum plasma concentration (Cmax) of futibatinib, binimetinib, and AR00426032 | approximately 24 months
  Plasma concentrations of futibatinib, binimetinib, and AR00426032
PK: Area under the plasma concentration-time curve (AUC) of futibatinib, binimetinib, and AR00426032 | approximately 24 months
  Plasma concentrations of futibatinib, binimetinib, and AR00426032
PK: Time to reach maximum plasma concentration (Tmax) of futibatinib, binimetinib, and AR00426032 | approximately 24 months
  Plasma concentrations of futibatinib, binimetinib, and AR00426032
PK: Terminal elimination half-life (T1/2) of futibatinib, binimetinib, and AR00426032 | approximately 24 months
  Plasma concentrations of futibatinib, binimetinib, and AR00426032
PK: Minimum plasma concentration before administration (Cmin) of futibatinib, binimetinib, and AR00426032 | approximately 24 months
  Plasma concentrations of futibatinib, binimetinib, and AR00426032
PK: Accumulation ratio of Cmax and AUC (R) of futibatinib, binimetinib, and AR00426032 | approximately 24 months
  Plasma concentrations of futibatinib, binimetinib, and AR00426032
Duration of response (DOR) | approximately 24 months
  DOR is defined as the length of time between first response and the date of objectively documented progression of disease or death
Progression-free survival (PFS) | approximately 24 months
  PFS is defined as the time from date of first dose to objectively documented progression of disease or death
Disease control rate (DCR) at 24 months | approximately 24 months
  DCR is defined as the percentage of patients who have achieved a CR, PR, or SD.
Number of patients with treatment-emergent adverse events as assessed by CTCAE v5.0 | Approximately 24 months
  Evaluate safety and tolerability of futibatinib in combination with binimetinib based on treatment-emergent adverse events per CTCAE v5.0(including serious adverse events),clinical laboratory parameters, ECGs, and vital signs

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of California Los Angeles UCLA Cancer, Santa Monica, California
  - Community Cancer Center North, Indianapolis, Indiana
  - The University of Texas MD Anderson Cancer Center, Houston, Texas